CLINICAL TRIAL: NCT00350610
Title: Computer-Based Training in Cognitive Behavior Therapy
Acronym: CBT4CBT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0207017894; DA015969
Record Dates: First submitted 2006-07-07; First posted 2006-07-11 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Cocaine Abuse
Keywords: cognitive behavior therapy; computer assisted instruction; drug abuse therapy; educational resource design and development
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Standard treatment as usual (TAU) in a community based clinic consisting of individual and group therapy sessions and regular urine monitoring.
  Interventions: Other: Treatment as usual (TAU)
- 2 (Experimental): Standard treatment as usual (TAU) plus coping skills computer program. In addition to the individual and group therapy sessions (TAU), individuals will work with a computerized program that teaches skills for stopping cocaine use and increasing coping skills twice weekly for 8 weeks.
  Interventions: Other: Treatment as usual (TAU); Behavioral: CBT for CBT

INTERVENTIONS:
Other: Treatment as usual (TAU) — Standard treatment as usual in a community based treatment setting
Behavioral: CBT for CBT — Standard treatment as usual (TAU) plus computer based therapy using CBT
  Arms: 2

SUMMARY:
The computer-based training program (CBT for CBT) focuses on teaching basic coping skills, presenting examples of effective use of coping skills in a number of realistic situations in video form, and providing opportunities for patients to practice and review new skills while receiving substance abuse treatment.

DETAILED DESCRIPTION:
In this behavioral trial 120 methadone maintained cocaine abusing individuals will be randomly assigned to either treatment as usual in a community-based clinic OR treatment as usual plus 8 hours of access to the 'CBT for CBT' computer program over a period of 8 weeks. Primary outcomes will be retention in treatment and reduction in cocaine use (percent days abstinent, confirmed by urine toxicology screens). The patients' ability to demonstrate coping skills through a computerized role-play evaluation will be a secondary outcome. A six-month follow-up will assess durability and/or delayed emergence of effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* methadone maintained for at least 3 months
* meet current DSM-IV criteria for cocaine use disorder
* fluent in English or at least a6th grade reading level
* can commit to at least 8 weeks of treatment and willing to be randomized to treatment

Exclusion Criteria:

* untreated bipolar or schizophrenic disorder
* current legal case pending (pending incarceration during 8 weeks of study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
reduction in drug use | 8 weeks

SECONDARY OUTCOMES:
patients ability to demonstrate coping skills through a computerized role-playing evaluation | 8 weeks
retention in treatment | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Carroll, PhD, Principal Investigator — Yale University/Department of Psychiatry
Locations (1):
- APT Foundation Orchard Hill Clinic, New Haven, Connecticut, United States

REFERENCES:
- [Derived] DeVito EE, Kober H, Carroll KM, Potenza MN. fMRI Stroop and behavioral treatment for cocaine-dependence: Preliminary findings in methadone-maintained individuals. Addict Behav. 2019 Feb;89:10-14. doi: 10.1016/j.addbeh.2018.09.005. Epub 2018 Sep 6. PMID 30240978
- [Derived] Decker SE, Morie K, Hunkele K, Babuscio T, Carroll KM. Emotion regulation strategies in individuals with cocaine use disorder maintained on methadone. Am J Addict. 2016 Oct;25(7):529-32. doi: 10.1111/ajad.12439. Epub 2016 Sep 22. PMID 27658192
- [Derived] Morie KP, Nich C, Hunkele K, Potenza MN, Carroll KM. Alexithymia level and response to computer-based training in cognitive behavioral therapy among cocaine-dependent methadone maintained individuals. Drug Alcohol Depend. 2015 Jul 1;152:157-63. doi: 10.1016/j.drugalcdep.2015.04.004. Epub 2015 Apr 27. PMID 25982006
- [Derived] Carroll KM, Kiluk BD, Nich C, Gordon MA, Portnoy GA, Marino DR, Ball SA. Computer-assisted delivery of cognitive-behavioral therapy: efficacy and durability of CBT4CBT among cocaine-dependent individuals maintained on methadone. Am J Psychiatry. 2014 Apr;171(4):436-44. doi: 10.1176/appi.ajp.2013.13070987. PMID 24577287
- [Derived] Worhunsky PD, Stevens MC, Carroll KM, Rounsaville BJ, Calhoun VD, Pearlson GD, Potenza MN. Functional brain networks associated with cognitive control, cocaine dependence, and treatment outcome. Psychol Addict Behav. 2013 Jun;27(2):477-88. doi: 10.1037/a0029092. Epub 2012 Jul 9. PMID 22775772
- [Derived] Carroll KM, Kiluk BD, Nich C, Babuscio TA, Brewer JA, Potenza MN, Ball SA, Martino S, Rounsaville BJ, Lejuez CW. Cognitive function and treatment response in a randomized clinical trial of computer-based training in cognitive-behavioral therapy. Subst Use Misuse. 2011;46(1):23-34. doi: 10.3109/10826084.2011.521069. PMID 21190403